CLINICAL TRIAL: NCT00932022
Title: Trospium Chloride XR in Obese Female Patients With Overactive Bladder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MA-SXR-09-003; Sanctura XR obesity OAB Trial (Other: Allergan)
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Results first posted 2013-01-21 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2012-12

CONDITIONS: Obesity; Overactive Bladder; Incontinence
MeSH Terms: conditions — Obesity; Urinary Bladder, Overactive | interventions — trospium chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- trospium chloride XR 60 mg (Experimental): Placebo capsule taken orally once daily for 2 weeks followed by trospium chloride extended release (XR) 60 mg capsule taken orally once daily for 12 weeks.
  Interventions: Drug: Trospium Chloride, Extended Release (XR); Other: placebo
- placebo (Placebo Comparator): Placebo capsule taken orally once daily for 14 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Trospium Chloride, Extended Release (XR) — Trospium chloride extended release 60 mg capsule taken orally once daily for 12 weeks.
  Other Names: Sanctura XR™ 60 mg
  Arms: trospium chloride XR 60 mg
Other: placebo — Placebo capsule taken orally once daily for either 2 weeks or 14 weeks.

SUMMARY:
This study evaluated the effectiveness of trospium chloride extended release (XR) in obese female patients with overactive bladder (OAB). Patients received either placebo and trospium chloride XR or placebo only. The study assessed the change from baseline in urinary frequency, urgency, and incontinence for trospium chloride XR versus a placebo-pill. The study was 14 weeks in duration.

ELIGIBILITY:
Inclusion Criteria:

* OAB syndrome with Urgency, Urinary frequency and Urgency urinary incontinence
* Non-smoker (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc., for 6 months prior to the screening visit).
* Obese

Exclusion Criteria:

* Chronic kidney failure
* Abdominal bypass surgery for obesity
* Moderate or severe memory impairment
* Uncontrolled narrow angle glaucoma
* Uncontrolled systemic disease
* Concurrent dementia drugs: Aricept (donepezil), Namenda (memantine), Cognex (tacrine), Exelon (rivastigmine), Razadyne (galantamine), or similar drugs for dementia

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- La Mesa, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trospium Chloride XR 60 mg | Placebo
Started | 64 | 63
Completed | 59 | 59
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trospium Chloride XR 60 mg | Placebo | Total
Number analyzed (Participants) | 64 | 63 | 127
Age, Customized [Number; unit: Participants]
  <18 years | 0 | 0 | 0
  18 to 75 years | 64 | 63 | 127
  >75 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 63 | 127
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Urinary Urgency Incontinence (UUI)
Description: Patients recorded information about UUI (accidental leakage, urgency associated with void and urgency severity) in a 3-day diary at Baseline (Week 2) and Week 14. The daily average episodes of UUI was the sum of all UUI episodes over valid diary days during the 3-day diary period divided by the valid number of diary days with at least one valid bladder entry. The percent change from baseline was calculated as (Mean UUI at Week 14- Mean UUI at Week 2)/ Mean UUI at Week 2 X 100. A negative number percent change from baseline indicated an improvement.
Time Frame: Baseline (Week 2), Week 14
Population: Modified Intent-to-Treat (mITT) defined as all patients who were randomized and received at least one dose of study medication. Analysis below was done on patients from the mITT population who completed the study at Week 14 and who had data available for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Trospium Chloride XR 60 mg | Placebo
Number analyzed (Participants) | 54 | 49
Percent change | -23.7 (36.16) [-88.9 to 50.0] | 57.8 (275.3) [-73.7 to 1400]

2. Secondary Outcome: Percent Change From Baseline in Urgency Severity Associated With Toilet Voids
Description: Due to lack of evaluable data, analysis for this outcome measure was not performed.
Time Frame: Baseline (Week 2), Week 14
Arm/Group | Trospium Chloride XR 60 mg | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percent Change From Baseline in Voided Volume
Description: Due to lack of evaluable data, analysis for this outcome measure was not performed.
Time Frame: Baseline (Week 2), Week 14
Arm/Group | Trospium Chloride XR 60 mg | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percent Change From Baseline in Over Active Bladder (OAB)-Symptom Composite Score
Description: Due to lack of evaluable data, analysis for this outcome measure was not performed.
Time Frame: Baseline (Week 2), Week 14
Arm/Group | Trospium Chloride XR 60 mg | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percent Change From Baseline in Percentage of Patients Continent
Description: Due to lack of evaluable data, analysis for this outcome measure was not performed.
Time Frame: Baseline (Week 2), Week 14
Arm/Group | Trospium Chloride XR 60 mg | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The safety population was used to calculate the number of participants at risk for Serious Adverse Events and Adverse Events and was defined as all randomized and treated participants.
Arm/Group | Trospium Chloride XR 60 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/64 | 1/63
Other Adverse Events (participants affected / at risk) | 6/64 | 3/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trospium Chloride XR 60 mg (N=64) | Placebo (N=63)
Atrial fibrillation (Cardiac disorders) | 0 | 1 — Event occurred prior to randomization to study medication.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trospium Chloride XR 60 mg (N=64) | Placebo (N=63)
Dry mouth (General disorders) | 6 | 3

LIMITATIONS AND CAVEATS:
Due to lack of evaluable data, analysis for the secondary outcome measures was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.